CLINICAL TRIAL: NCT05832372
Title: Esophagogastric Histopathology Potentially Guided Patients Younger Than 50 Years Old to Undergo Colonoscopy Earlier: A Retrospective Cross-sectional Study
Brief Title: Esophagogastric Histopathology Potentially Guided Patients Younger Than 50 Years Old to Undergo Colonoscopy Earlier
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Clinical Professor, Shandong University
Other Study IDs: 2023033
Record Dates: First submitted 2023-03-27; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal colonoscopy group: Individuals with normal colonoscopy examination
- Colorectal polyps group: Individuals with colorectal polyps diagnosed by colonoscopy

SUMMARY:
Colorectal cancer (CRC) is the third most diagnosed cancer worldwide and second leading cause of cancer death. Most CRCs arise from a polyp, developing through two major precursor lesion pathways: the traditional adenoma-carcinoma pathway, and the serrated neoplasia pathway. This provides opportunities to prevent cancer by removing its precursor lesions. CRC screening efforts are directed toward removal of precancerous polyps with colonoscopy and detection of early-stage CRC, which has been demonstrated to reduce CRC incidence and mortality effectively, making CRC one of the most preventable and treatable forms of cancer.

Current guidelines in China recommend starting CRC screening uniformly at age 50 in average-risk individuals. However, a one-fits-all approach to determining CRC screening starting age may be not conducive to personalized screening, especially in the developing countries with scarce health resources. The incidence of early-onset CRC (CRC diagnosed before the age of 50) has shown a continuous increasing trend worldwide, spurring the US Preventive Services Task Force to recommend initiating average-risk CRC screening at age 45 instead of 50. Furthermore, different populations may benefit from even earlier screening, and CRC incidence may differ on the basis of population characteristics and CRC risk factors. For individuals younger than 50 years old, earlier screening based on risk factors may address this concern.

Previous studies have recommended earlier starting age of CRC screening combined with risk factors such as but not limited to sex, age, family history, lifestyle and comorbidity. Some upper gastrointestinal diseases have also been reported to be associated with an increased risk of colorectal neoplasms, which may be related to the destruction of gastric acid barrier function and long-term use of pump proton inhibitors. Compared with colonoscopy examination, individuals were more willing to undergo esophagogastroduodenoscopy (EGD) examination for gastric cancer screening, especially among the younger, potentially utilizing the EGD to guide earlier colonoscopies for patients at increased risk. Therefore, this study was aimed to investigate the association between esophagogastric histopathology and colorectal neoplasms in patients under the age of 50 and whether these risks factor could be combined with to guide earlier CRC screening.

ELIGIBILITY:
Inclusion Criteria:

Patients younger than 50 years old who underwent gastroscopy and colonoscopy simultaneously.

Exclusion Criteria:

1. Patients without a good bowel preparation (Boston Bowel Preparation Scale [BBPS] score ≥ 6);
2. Incomplete gastroscopy or colonoscopy examinations;
3. Partial or total gastrointestinal resection;
4. Patients who have been diagnosed with gastrointestinal cancer before endoscopy;
5. Hereditary polyposis, including Peutz-Jeghers syndrome, and familial adenomatous polyposis;
6. A history of inflammatory bowel diseases.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This retrospective observational study analyzed records between November 7, 2020, and November 14, 2022 which were extracted from Qilu Hospital of Shandong University. Patients younger than 50 years old who underwent gastroscopy and colonoscopy simultaneously, were selected and enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-05-27 (Estimated); Study Completion 2023-05-27 (Estimated)

PRIMARY OUTCOMES:
Prevalence or occurrence of upper gastrointestinal diseases | 1 year
  Including Helicobacter pylori, atrophic gastritis/intestinal metaplasia, reflux esophagitis, Barrett's esophagus, peptic ulcer, gastric polyps, low-grade intraepithelial neoplasia (LGIN), and high-grade intraepithelial neoplasia (HGIN).